CLINICAL TRIAL: NCT02160886
Title: Effects of a Task Oriented Intervention for Children With Disabilities, Based on Children's or Parent's Goals, a Randomized Study.
Brief Title: Effects of a Task Oriented Intervention With Two Goal-setting Approaches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Gävleborg (Other)
Responsible Party: Principal Investigator, Kristina Vroland Nordstrand, PhD-student, Region Gävleborg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RFR-296311
Record Dates: First submitted 2014-06-08; First posted 2014-06-11 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Movement Disorder; Learning Disability; Autism Spectrum Disorder; Children
MeSH Terms: conditions — Movement Disorders; Learning Disabilities; Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Child-goal (Experimental): The children will receive goal- directed task oriented interventions based on goals identified by the children themselves, using the Swedish version of the Perceived Efficacy and Goal Setting System (PEGS).
  A PEGS interview will be performed with the children. The children identifies tasks they find difficult to perform and prioritize three tasks, they want to perform better, as goals for intervention.
  Interventions: Behavioral: child-goal
- Parent-goal (Experimental): The children will receive goal- directed task oriented interventions based on goals identified by the parents using the Canadian Occupational Performance Measure (COPM).
  Using the COPM interview technique, the parents are encouraged to talk about an ordinary day to identify occupational performance issues their child is not able to perform. Identified performance issues are rated for importance and the parents selects the three most important issues as goals for intervention.
  Interventions: Behavioral: parent-goal

INTERVENTIONS:
Behavioral: child-goal — The 8-week goal-directed intervention include completing a daily home program and a weekly follow-up session with the child's occupational therapist.
  The parents are responsible for the day to day practice and are encouraged to let the children practice daily in their natural environment.
  The home-programs focus on enhancing the agreed upon goal specific task performance. They include structured practice of tasks and adaptations and modifications of the environment and the tasks.
  The weekly sessions with the occupational therapist are meant to sustain motivation, follow-up on progress, adjust the home program for the coming week and support parents in how to carry out the daily interventions.
  Arms: Child-goal
Behavioral: parent-goal — The 8-week goal-directed intervention include completing a daily home program and a weekly follow-up session with the child's occupational therapist.
  The parents are responsible for the day to day practice and are encouraged to let the children practice daily in their natural environment.
  The home-programs focus on enhancing the agreed upon goal specific task performance. They include structured practice of tasks and adaptations and modifications of the environment and the tasks. .
  The weekly sessions with the occupational therapist are meant to sustain motivation, follow-up on progress, adjust the home program for the coming week and support parents in how to carry out the daily interventions.
  Arms: Parent-goal

SUMMARY:
A randomized trial investigating if effects of a goal-directed task oriented intervention is influenced by who takes the decision and establishes the goal (the child or the parent) and whether establishing a goal per se influence performance and goal-achievement. The main hypothesis are that children's participation in the goal-setting process would positively influence goal achievement, children's self-identified goals would be achievable and that both groups would achieve goals that were the target of a goal-directed intervention.

ELIGIBILITY:
Inclusion Criteria:

* enrollment in pediatric rehabilitation, age between 5-12 years and any type of disability but functioning at or above a 5 year old level in receptive language.

Exclusion Criteria:

* involvement in another block of intensive intervention during the 5-month study period

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2011-10; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Goal Attainment Scaling (GAS) | Three times, at baseline, post-intervention (8-weeks) and follow-up (5-months)
  The purpose of the Goal Attainment Scaling, GAS is to measure goal attainment. GAS is an individualized criterion-referenced measure it involves describing current performance and specifying a range of outcomes for a specific goal, using the scale to evaluate the individual change after a specific intervention period

SECONDARY OUTCOMES:
Performance scale of the Canadian Occupational Performance Measure | Assesed once a week up to 11 weeks which include three baseline assesments and eight assesments during the egiht weeks intervention period
  The performance scale of the Canadian Occupational Performance Measure is a 10 point rating scale of ability of performance of a specific task, the purpose is to detect change in an individual's perception of the occupational performance.
Beck Youth scales, subscale self-concept | Three times, at baseline, post-intervention (eigth weeks) and at follow-up (5-months)
  The purpose of the subscale self-concept in the Beck Youth Scales is to measures the child's estimated perceived self-concept.

OTHER OUTCOMES:
Pediatric Evaluation of Disability Inventory (PEDI) | One time, at baseline
  The purpose of the Caregiver assistance scale of the PEDI, is to describes children's need for assistance in everyday tasks within the domains of self-care, mobility and social function.
Parental questionnaire | Assesed once a week up to egiht weeks during the eight weeks intervention period
  The purpose of the parental questionnaire developed for the study is to capture the parents' perception of the coaching burden and motivation to practice at home.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Vroland-Nordstrand, Phd-student, Principal Investigator — Department of Women's and Children's Health Karolinska Institutet; Lena Krumlinde-Sundholm, Assoc Prof, Principal Investigator — Department of women's and Children's Helath Karolinska Institutet; Ann-Christin Eliasson, Professor, Principal Investigator — Department of women's and children's Health, Karolinska Institutet
Locations (1):
- Gävleborg County Council, Gävle, Sweden